CLINICAL TRIAL: NCT04053543
Title: A Phase 2, Multi-Center, Open-Label Study to Evaluate Long-term Safety and Efficacy of CXA-10 in Subjects With Pulmonary Arterial Hypertension on Stable Background Therapy: Extension to Study CXA-10-301
Brief Title: CXA-10 Study in Subjects With Pulmonary Arterial Hypertension
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: LOE
Sponsor: Complexa, Inc. (Industry)
Collaborators: Medpace, Inc. (Industry); Innovative Analytics (Unknown); Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CXA-10-2302
Record Dates: First submitted 2019-07-19; First posted 2019-08-12 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: PAH
Keywords: Pulmonary Arterial Hypertension; Pulmonary Hypertension; PAH; Connective Tissue Disease- Associated; 6 Minute Walk Test; 6 Minute Walk Distance; Pulmonary Vascular Resistance; Cardiac MRI; Right Ventricular Function; Hypertension; Familial Primary Pulmonary Hypertension; Connective Tissue Diseases; Vascular Diseases; Hypertension, Pulmonary; Lung Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary; Hypertension; Familial Primary Pulmonary Hypertension; Connective Tissue Diseases; Vascular Diseases; Lung Diseases; Cardiovascular Diseases | interventions — CXA-10

STUDY DESIGN:
Intervention Model Description: CXA-10
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 150mg CXA-10 (Experimental): Once daily dosing of 150mg CXA-10 in the morning
  Interventions: Drug: CXA-10

INTERVENTIONS:
Drug: CXA-10 — (10-nitro-9(E)-octadec-9enoic acid)

SUMMARY:
This is a Phase 2, multicenter, open-label extension (OLE) of study CXA-10-301, to evaluate the long term safety and efficacy of daily dosing of CXA-10.

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, open-label extension (OLE) of study CXA-10-301, to evaluate the long term safety and efficacy of daily dosing of CXA-10.

The study will be performed in approximately 50 study centers across the United States and the United Kingdom, which participated in CXA-10-301. Approximately 96 subjects who completed treatment in CXA-10-301 will be eligible to participate in this OLE study, after completing all Visit 9 (Day 1 and Day 2) assessments in CXA-10-301.

Study participation for each subject will last up to approximately 6.5 months. The study will consist of a 6 month open-label treatment period and require 5 clinic visits and 1 telephone visit, including the Baseline Visit completed simultaneously with Visit 9 CXA-10-301, plus a follow-up visit approximately 2 weeks following the last dose of CXA-10.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document indicating subject has been informed of all pertinent aspects of the study prior to initiation of any study-required procedures.
2. Is willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.
3. Has completed the CXA-10-301 study and demonstrated compliance with study medication administration and study requirements.
4. If receiving simvastatin-containing products: simvastatin (Zocor), Vytorin, or any other combination therapy containing simvastatin, simvastatin dose does not exceed 20 mg/day.
5. Currently receiving no more than three of the following previously approved PAH therapies: phosphodiesterase type 5 (PDE-5) inhibitors, endothelin receptor antagonists (ERA), soluble guanylate cyclase (sGC) stimulator, prostanoids, prostacyclin receptor agonists.
6. Women of childbearing potential and males with partners of childbearing potential must agree to use a reliable method of contraception while taking study medication.

Exclusion Criteria:

1. Severe hypotension defined by systolic blood pressure <90 mmHg from sitting blood pressure measurement at Baseline.
2. Hypertensive defined by >160 mmHg systolic or >110 mmHg diastolic from sitting blood pressure measurement at Baseline.
3. QTcF on supine ECGs at Baseline (Visit 1) of >500 msec.
4. Acute myocardial infarction or acute coronary syndrome (ST-Elevation Myocardial Infarction [STEMI], Non STEMI [NSTEMI] and or unstable angina) within the last 90 days prior to Baseline.
5. Recent cerebrovascular accident/transient ischemic attack (CVA/TIA) within the last 90 days prior to Baseline.
6. Recent hospitalization for left heart failure within the last 90 days prior to Baseline.
7. Clinically significant aortic or mitral valve disease defined as greater than mild regurgitation or mild stenosis; pericardial constriction; restrictive or constrictive cardiomyopathy; left ventricular dysfunction (LVEF < 50%); left ventricular outflow obstruction; symptomatic coronary artery disease; autonomic hypotension; or fluid depletion, in the opinion of the investigator.
8. Chronic atrial fibrillation and life-threatening cardiac arrhythmias.
9. Personal or family history of congenital prolonged QTc syndrome or sudden unexpected death due to a cardiac reason.
10. Clinically significant anemia in the opinion of the investigator that precludes enrollment into this study, or Hb <9 gm/dl.
11. Severe hepatic impairment (Child-Pugh class C with or without cirrhosis) at Baseline or active chronic hepatitis.
12. Received intravenous inotropes within 2 weeks prior to Baseline (e.g. dopamine, dobutamine).
13. History of angina pectoris or other condition that was treated with long or short acting nitrates <12 weeks of Baseline.
14. History of herbal or natural medication use (including fish oil) within 2 weeks or 5 half-lives, whichever is longer, prior to Baseline.
15. Received prednisone at doses > 15 mg/ day or changes in immunosuppressive medications <12 weeks prior to Baseline.
16. Currently taking a drug that may affect the assay measurement of serum creatinine (e.g. cimetidine, Bactrim, Pyridium). A list is provided in Appendix H.

21. Newly prescribed drug or increased dose of an existing drug that is known to prolong the QTc interval and has been associated with Torsades de Pointes (TdP) identified in the CredibleMeds.org website list as known risk (KR) of TdP.

Note: Stable doses of drugs classified as conditional risk (CR) of TdP or possible risk (PR) of TdP are permitted (i.e., subject has received the same dose and regimen for at least 30 days prior to Baseline with no anticipated changes to the dose or regimen during the course of the study).

22. Currently taking dimethyl fumarate (Tecfidera™).

23. Any of the following laboratories abnormal and unresolved in CXA-10-301:

1. Absolute lymphocyte counts < 0.5 x 109 cells/L.
2. Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 3.0X upper limit of normal (ULN), alkaline phosphatase (AP) > 2X ULN of liver origin, and total bilirubin >2X ULN. If all liver function tests (LFTs) are within normal limits (WNL) and total bilirubin is elevated, examination of direct and indirect bilirubin may be conducted to evaluate for Rotor's/Gilbert's Syndrome. Subjects with Rotor's/Gilbert's Syndrome may be enrolled.
3. eGFR < 30 mL/min/1.73 m2 (estimated by Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] Creatinine/Cystatin C 2012 algorithm) at Baseline.

   24. Females who are pregnant or breastfeeding, or who are trying to conceive. 25. Recent (within 1 year) history of abusing alcohol or illicit drugs. 26. History of any primary malignancy, including a history of melanoma or suspicious undiagnosed skin lesions, or other malignancies (such as thyroid or testicular) that have been curatively treated and with no evidence of disease for at least 3 years or prostate cancer who is not currently or expected, during the study, to undergo radiation therapy, chemotherapy, and/or surgical intervention, or to initiate hormonal treatment.

   Exception: subjects with history of basal cell or squamous cell carcinomas of the skin or cervical carcinoma in situ are eligible for enrollment.

   27. Cardiovascular, liver, renal, hematologic, gastrointestinal, immunologic, endocrine, metabolic, central nervous system or psychiatric disease that, in the opinion of the investigator, may adversely affect the safety of the subject and/or efficacy of the investigational product or severely limit the lifespan of the subject other than the condition being studied.

   28. Clinically significant hyperthyroidism or hypothyroidism not adequately treated.

   29. Any other condition and/or situation that causes the Investigator to deem a subject unsuitable for the study (e.g., due to expected study medication non- compliance, inability to medically tolerate the study procedures, or a subject's unwillingness to comply with study-related procedures).

   30. Known hypersensitivity to CXA-10, the metabolites, or formulation excipients.

   31. Treatment with any investigational drug (other than CXA-10) or device within 30 days or 5 half-lives (whichever is longer) prior to Baseline (this includes investigational formulations of marketed products, inhaled and topical drugs), or plans to participate in an investigational drug or device study at any time during this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2020-08-12 (Actual)

PRIMARY OUTCOMES:
Incidence of AEs | 6 months
  Adverse events occurring during the treatment period
Changes in respiration | 6 months
  Change from baseline values at each post-baseline time point
Changes in heart rate | 6 months
  Change from baseline values at each post-baseline time point
Changes in blood pressure | 6 months
  Change from baseline values at each post-baseline time point

SECONDARY OUTCOMES:
PAH-specific medication changes | 6 months
  Addition or removal of PAH-specific medications, including any dose changes
6 Minute Walk Distance | 6 months
  Change from baseline in 6-minute walk distance (6MWD)
Who Classification of Functional Status | 6 months
  Change from baseline in WHO Classification of Functional Status of Patients with PH
Clinical worsening | 6 months
  Death from any cause, hospitalization for worsening PAH, Disease progression, unsatisfactory long-term clinical response

CONTACTS AND LOCATIONS:
Overall Officials: Theo Danoff, MD, Study Director — Complexa, Inc.
Locations (37):
- United States (31):
  - University of Alabama, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - University of California San Diego, La Jolla, California
  - University of California San Francisco, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - Washington Hospital (Medstar), Washington D.C., District of Columbia
  - George Washington Medical Faculty Associates, Washington D.C., District of Columbia
  - University of Florida Health, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Kansas, Kansas City, Kansas
  - University of Minnesotta, Minneapolis, Minnesota
  - Washington University and Barnes Jewish Hospital, St Louis, Missouri
  - NYU Langone Medical Center, New York, New York
  - Duke University, Durham, North Carolina
  - Christ Hospital-Lindner Research Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Vanderbuilt University, Nashville, Tennessee
  - UT Southwestern, Dallas, Texas
  - Texas Tech, El Paso, Texas
  - Houston Methodist, Houston, Texas
  - University of Virginia School of Medicine, Charlottesville, Virginia
  - Inova Medical Campus, Falls Church, Virginia
  - Sentara Medical Group, Norfolk, Virginia
  - Froedert Medical College of Wisconsin, Milwaukee, Wisconsin
- United Kingdom (6):
  - Golden Jubilee National Hospital, Glasgow
  - Royal Free, London
  - Royal Brompton, London
  - Hammersmith Hospital, London
  - Freeman Hospital, Newcastle upon Tyne
  - Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Undecided